CLINICAL TRIAL: NCT06232798
Title: A Single-Center, Exploratory Clinical Study Combining Radiofrequency and Pulsed Field Ablation for Persistent Atrial Fibrillation Based on Columbus™ 3D EP Navigation System
Brief Title: A Dual Energy Catheter (PFA and RFA) and a PFA Catheter for the Treatment of PeAF
Acronym: PFA，RFA，PeAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort EP MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 775046
Record Dates: First submitted 2024-01-18; First posted 2024-01-31 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Persistent Atrial Fibrillation
Keywords: PFA; PeAF; PFA/RF
MeSH Terms: conditions — Atrial Fibrillation | interventions — Desmoglein 1; Catheter Ablation; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: A prospective, singelcenter, single-arm clinical study to evaluate the safety and efficacy of PFA/RF catheter or PFA catheter for the treatment of persistent atrial fibrillation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A prospective, singlecenter, single-arm clinical study (Experimental)
  Interventions: Other: a dual energy catheter (RF and PFA) or PFA catheter only will be to treat PeAF,Cardiac Pulsed Electric Field Ablation Catheter; Other: catheter ablation

INTERVENTIONS:
Other: a dual energy catheter (RF and PFA) or PFA catheter only will be to treat PeAF,Cardiac Pulsed Electric Field Ablation Catheter — This study will be used two catheters, the contact force sensing catheter able to deliver both RF and PFA energy, this catheter provides both the radiofrequency (RF) energy and pulsed field ablation (PFA) energy to the catheter through the toggling of the two energy sources on the generator monitor. Another catheter is PFA catheter only.
Other: catheter ablation — catheter ablation
  Other Names: operation

SUMMARY:
The goal of this clinical trial is to treatment of patients with persistent atrial fibrillation with PFA/RFA. 10 patients will be treated by PFA/RFA catheter or PFA catheter only.

Participants will followed 1、3 month after catheter ablation

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old;
2. Documented symptomatic persistent atrial fibrillation, defined as persistent atrial fibrillation lasting more than 7 days and less than 1 year；
3. Ineffective or intolerable after treatment with at least one Class I or Class III antiarrhythmic drug;
4. Fully understand the treatment protocol and voluntarily sign the informed consent form and be willing to undergo the tests, procedures and follow-ups required by the protocol.

Exclusion Criteria:

1. Patients who have undergone left atrial surgery
2. Left atrial thrombosis
3. Patients with combined atrial tachycardia and atypical atrial flutter
4. Patients of childbearing age who are unable to use effective contraception during the 3-month period following enrollment
5. Anterior and posterior left atrial diameter ≥ 55mm
6. Left ventricular ejection fraction (LVEF) ≤ 40%
7. Previous atrial septal repair or atrial mucinous tumor
8. Active implants (e.g. pacemakers, ICDs, etc.) in the body
9. NYHA class III-IV cardiac function
10. Clear cerebrovascular disease within the last 6 months (including cerebral hemorrhage, stroke, transient ischemic attack)
11. Cardiovascular events within the last 3 months (including acute myocardial infarction, coronary intervention or heart bypass surgery, prosthetic valve replacement or repair, atrial or ventriculotomy)
12. Those with acute or severe systemic infections
13. Patients with severe liver or kidney disease, malignant tumors or end-stage disease that, in the opinion of the investigator, may interfere with the treatment, evaluation and compliance of this trial
14. Patients with significant bleeding tendency, hypercoagulable state and severe hematologic disorders
15. Patients who have participated or are participating in other clinical trials within 3 months prior to enrollment
16. Patients who have other conditions that the investigator considers inappropriate for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Immediate success rate | 1 Day of catheter ablation
  Refers to the proportion of the number of subjects electrically isolated in each AF patient after surgery to the total number of subjects enrolled.

SECONDARY OUTCOMES:
Ablation success at 3-month after the catheter ablation | 3 months
  Ablation success is defined as no recurrence with no anti-arrhythmic drugs by taking history of symptoms from the patient and by Holter 24 Hours.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China